CLINICAL TRIAL: NCT01327794
Title: The Relationship of Serum 25-Hydroxyvitamin D to Overall Survival in Advanced Pancreatic Cancer
Brief Title: Relationship Between Vitamin D Biomarkers and Survival in Blood Samples From Patients With Advanced Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151006; U10CA031946 (NIH); CALGB-151006; CDR0000698059 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis; Immunologic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Participants in this correlative study (CALGB 151006) were enrolled in CALGB 80303, which was a national, multi-center, double-blind phase III study that randomly assigned patients (1:1) with advanced pancreatic cancer to gemcitabine plus bevacizumab vs gemcitabine plus placebo. Blood samples were collected from consenting participants in CALGB 80303 at the time of study registration at respective institutions and shipped to the CALGB Pathology Coordinating Office for storage (Columbus, OH).Baseline serum 25-hydroxyvitamin D (25[OH]D) levels were measured and examined associations between baseline 25(OH)D levels and progression-free survival and OS using the Cox rank score test.
  Interventions: Genetic: polymorphism analysis; Other: immunologic technique; Other: laboratory biomarker analysis; Other: medical chart review

INTERVENTIONS:
Genetic: polymorphism analysis
Other: immunologic technique
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research trial is studying the relationship between vitamin D biomarkers and survival in blood samples from patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective

* To measure baseline serum 25-hydroxyvitamin D (25[OH]D) levels in a cohort of patients with advanced pancreatic cancer enrolled in the Cancer and Leukemia Group B (CALGB) study 80303 and evaluate the association between vitamin D status and overall survival (OS) or progression free survival (PFS).

Secondary Objective

* To evaluate the association between common germ-line single nucleotide polymorphisms (SNPs) in the vitamin D pathway genes and 25(OH)D levels in patients with advanced pancreatic cancer.
* To evaluate the interaction between serum 25(OH)D levels and germ-line SNPs in the vitamin D pathway genes in predicting OS in advanced pancreatic cancer.

OUTLINE: This is a multicenter study.

Archived serum samples are analyzed for 25-hydroxyvitamin D levels by competitive chemiluminescence immunoassay. Results are then compared with the germ-line single nucleotide polymorphisms from the Genome-Wide Association Study (GWAS) and patients' clinical data.

ELIGIBILITY:
1. Eligible patients had unresectable adenocarcinoma of the pancreas
2. Received no prior therapy for metastatic disease (prior radiation and/or chemotherapy in the adjuvant setting were allowed).
3. Baseline Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. Adequate renal, liver, and bone marrow function were required.
5. Patients signed informed consent for participation in the therapeutic trial and consented to the companion study for biomarker research (CALGB-151006).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had unresectable adenocarcinoma of the pancreas and had received no prior therapy for metastatic disease (prior radiation and/or chemotherapy in the adjuvant setting were allowed).
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Association between 25(OH)D level and OS | 35 months post-randomization

SECONDARY OUTCOMES:
Association between 25(OH)D level and PFS | 25 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alan Venook, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York, United States